CLINICAL TRIAL: NCT06483763
Title: Evaluating the Impact of a Photoaging App Versus School-Based Educational Intervention on Adolescents' Knowledge, and Attitudes Towards Tobacco Use in Omani Public Schools: A Cluster Randomized Trial
Brief Title: Evaluating the Impact of a Photoaging App Versus School-Based Educational Intervention on Adolescents' Knowledge, and Attitudes Towards Tobacco Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Al Mahrouqi, Principal Investigator, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NU/COMHS/EBC005/2023
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Use Cessation; Smoking Cessation; Smoking Prevention
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation | interventions — Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group using the SmokerFace App from the Education Against Tobacco (EAT) program (Other): Trained medical students will deliver the intervention and will be conducted in the specific classrooms of enrolled schools. The school students will be taught how to use the SmokerFace App from the Education Against Tobacco (EAT) program (26) with parental supervision at home. Medical Students will send the links to download the app from the App Store (iOS) and Play Store (Android), along with an explanation of how to install and use the app.
  Interventions: Other: SmokerFace App from the Education Against Tobacco (EAT) program
- The group receiving of standardized school-based educational module (Other): The control arm will receive a standardized school-based educational module that aligns with the tobacco health hazards awareness educational toolkit provided by the World Health Organization.
  Interventions: Other: The use of standardized school-based educational module

INTERVENTIONS:
Other: SmokerFace App from the Education Against Tobacco (EAT) program — The SmokerFace App utilizes photo-aging technology that requires users to take a selfie. This selfie is processed by the software to generate four images depicting the consequences of smoking (or not smoking) one pack a day over both a one-year and 15 years. The app provides explanations of these smoking beauty-reducing visual outcomes and educates users about the aesthetic impacts of smoking, along with potential health consequences.
  Arms: The group using the SmokerFace App from the Education Against Tobacco (EAT) program
Other: The use of standardized school-based educational module — This module is designed to promote a tobacco- and nicotine-free environment and is validated by at least three experts in related fields (27). The intervention will be customized to fit the Omani sociocultural context and will be administered in the classrooms of respective schools by the same team of trained medical students
  Arms: The group receiving of standardized school-based educational module

SUMMARY:
Tobacco use is a leading cause of preventable morbidity and mortality worldwide. It has been estimated that by 2030, tobacco use will cause approximately 10 million deaths per year worldwide, with 70% of those occurring in low- and middle-income countries. Oman, a country in the Arabian Peninsula, is not immune to this global health problem. Tobacco use is prevalent among young people in Oman, and efforts to prevent and control tobacco use among youth are a public health priority.

This study employs a cluster randomized controlled trial design to assess the impact of a photo-gaining app versus a structured educational intervention on tobacco knowledge and attitudes among adolescents in Sohar, Oman. Boys' public schools serve as clusters, with students in grades 9 to 12 as participants. Schools are randomly assigned to either an intervention or control group. The intervention, facilitated by medical students trained at a local university, involves using the SmokerFace App to demonstrate the effects of smoking via photo-aging technology. The control group receives a standardized educational module endorsed by the World Health Organization. Primary outcomes focus on comparing tobacco knowledge levels between groups, while secondary outcomes examine attitudes towards tobacco use. Pre-intervention and post-intervention assessments are conducted using the modified WHO Global Youth Tobacco Survey. Randomization is implemented in two stages to ensure balance, and efforts are made to maintain blinding among outcome assessors and data analysts.

The proposed study is a cluster randomized trial aimed at evaluating the impact of a photo-aging app versus structured educational intervention on knowledge and attitude towards tobacco use and tobacco consumption habits among Omani adolescents. The results of this study will be important for developing effective strategies for preventing tobacco use among youth in Oman and other countries with similar socio-cultural contexts.

ELIGIBILITY:
Inclusion and Exclusions Criteria:

All Boys' public schools in Sohar, North Al-Batinah Region, from classes 9 to 12, were included in the study. Girls' schools as well as parents and students who declined participation were excluded from the study.

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 227 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The difference in the level of knowledge regarding the harmful effects of tobacco use between the intervention and control groups using the GYTS Scale | 12 Weeks

SECONDARY OUTCOMES:
The difference in the attitudes towards tobacco use between the intervention and control groups using the GYTS Scale | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Science and Technology, Sohar, Oman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Mahrouqi T, Al-Ghailani F, Al-Maqbali M, Al Saidi M, Prashanth GP. A cluster randomized trial comparing photoaging app and school based educational intervention for tobacco use prevention in adolescents. Sci Rep. 2025 May 2;15(1):15374. doi: 10.1038/s41598-025-00165-5. PMID 40316573